CLINICAL TRIAL: NCT00002462
Title: Phase III Randomized Trial of Adjuvant Involved-Field Radiotherapy vs No Adjuvant Therapy Following Remission Induction With MOPP/ABV Hybrid Chemotherapy in Patients With Stage III/IV Hodgkin's Disease
Brief Title: RT or No RT Following Chemotherapy in Treating Patients With Stage III/IV Hodgkin's Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-20884; EORTC-20884 (Other: EORTC)
Record Dates: First submitted 1999-11-01; First posted 2004-07-26 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Doxorubicin; Mechlorethamine; Prednisone; Procarbazine; Vinblastine; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: doxorubicin hydrochloride
Drug: mechlorethamine hydrochloride
Drug: prednisone
Drug: procarbazine hydrochloride
Drug: vinblastine sulfate
Drug: vincristine sulfate
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET photon therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with combination chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with no radiation therapy following chemotherapy in treating patients with stage III or stage IV Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare relapse-free survival and overall survival of patients with Stage III/IV Hodgkin's disease randomly assigned to adjuvant involved-field radiotherapy vs. no adjuvant therapy following remission induction with MOPP/ABV (nitrogen mustard/vincristine/procarbazine/prednisone/doxorubicin/bleomycin/vinblastine). II. Evaluate the therapeutic efficacy of MOPP/ABV hybrid chemotherapy in advanced Hodgkin's disease. III. Evaluate the prognostic significance of an early response to MOPP/ABV in patients with advanced Hodgkin's disease.

OUTLINE: Study randomized for adjuvant radiotherapy. All patients receive Induction chemotherapy on Regimen A, following which those in CR are randomized on Arms I and II. Regimen A: 7-Drug Combination Chemotherapy. MOPP/ABV Hybrid. Mechlorethamine, NM, NSC-762; Vincristine, VCR, NSC-67574; Procarbazine, PCB, NSC-77213; Prednisone, PRED, NSC-10023; Doxorubicin, DOX, NSC-123127; Bleomycin, BLEO, NSC-125066; Vinblastine, VBL, NSC-49842. Arm I: Radiotherapy. Involved-field irradiation using megavoltage equipment. Arm II: No further therapy.

PROJECTED ACCRUAL: 321 evaluable patients will be required; an annual accrual rate of 80 patients is anticipated.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven clinical or pathological Stage III/IV Hodgkin's disease Pathological Stage IIIAS disease with the spleen as the only site of subdiaphragmatic involvement excluded

PATIENT CHARACTERISTICS: Age: 15 to 70 Performance status: Not specified Life expectancy: No severe limits on life expectancy due to nonmalignant disease Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No severe cardiac disease that would preclude protocol therapy Pulmonary: No severe pulmonary disease that would preclude protocol therapy Other: No severe metabolic or neurologic disease that would preclude protocol therapy No concomitant or previous second malignancy except: Nonmelanomatous skin cancer In situ carcinoma of the cervix

PRIOR CONCURRENT THERAPY: No prior therapy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 1989-09 (Actual); Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Benefit of adjuvant involved field RT after entering complete remission with MOPP/ABV hybrid CT
Efficacy of MOPP/ABV hybrid CT

SECONDARY OUTCOMES:
Relapse free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John Raemaekers, MD, PhD, Study Chair — Universitair Medisch Centrum St. Radboud - Nijmegen
Locations (56):
- Belgium (9):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Hopital Universitaire Erasme, Brussels
  - C.H.U. Saint-Pierre, Brussels (Bruxelles)
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Centre Hospitalier Universitaire Brugmann, Brussels (Bruxelles)
  - Centre Hospitalier Universitaire de Tivoli, La Louvière
  - U.Z. Gasthuisberg, Leuven
  - U.Z. Sint-Rafael, Leuven
- National Cancer Institute of Egypt, Cairo, Egypt
- France (17):
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier General, Compiègne
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hotel Dieu de Paris, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - Hopital Jules Courmont - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Medico-Chirurgical Foch, Suresnes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Zentralkrankenhaus, Bremen, Germany
- Italy (2):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Dipartimente di Oncologia di Torino, Turin (Torino)
- Netherlands (19):
  - Leyenburg Ziekenhuis, 's-Gravenhage (Den Haag, the Hague)
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Integraal Kankercentrum Amsterdam, Amsterdam
  - Slotervaart Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Streekziekenhuizen Gooi-Noord, Blaricum
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - De Wever Ziekenhuis, Heerlen
  - Radiotherapeutisch Instituut, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Integraal Kankercentrum West, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Radboud University Hospital, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Rotterdam Cancer Institute, Rotterdam
  - Sophia Ziekehuis, Zwolle
- Poland (3):
  - Maritime Hospital, Gdynia
  - Jagiellonian University, Krakow (Cracow)
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (3):
  - Hospitais da Universidade de Coimbra (HUC), Coimbra
  - Instituto Portugues de Oncologia de Francisco Gentil, Lisbon
  - Instituto Portugues de Oncologia do Porto, Porto
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Result] Aleman BM, Raemaekers JM, Tomisic R, Baaijens MH, Bortolus R, Lybeert ML, van der Maazen RW, Girinsky T, Demeestere G, Lugtenburg P, Lievens Y, de Jong D, Pinna A, Henry-Amar M; European Organization for Research and Treatment of Cancer (EORTC) Lymphoma Group. Involved-field radiotherapy for patients in partial remission after chemotherapy for advanced Hodgkin's lymphoma. Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):19-30. doi: 10.1016/j.ijrobp.2006.08.041. Epub 2006 Nov 9. PMID 17097834
- [Result] Aleman BM, Girinsky T, van der Maazen RW, Strijk S, Meijnders P, Bortolus R, Olofsen-van Acht MJ, Lybeert ML, Lievens Y, Eghbali H, Noordijk EM, Tomsic R, Meerwaldt JH, Poortmans PM, Smit WG, Pinna A, Henry-Amar M, Raemaekers JM; European Organization for Research; Treatment of Cancer (EORTC) Lymphoma Group. Quality control of involved-field radiotherapy in patients with advanced Hodgkin's lymphoma (EORTC 20884). Int J Radiat Oncol Biol Phys. 2005 Nov 15;63(4):1184-90. doi: 10.1016/j.ijrobp.2005.03.044. Epub 2005 Jun 2. PMID 15936157
- [Result] Aleman BMP, Girinsky T, Strijk S, et al.: Quality control of involved-field radiotherapy in patients with advanced stage Hodgkin's lymphoma (HL) enrolled on the EORTC trial 20884. [Abstract] Eur J Haematol 73 (Suppl 65): A-A02, 42, 2004.
- [Result] Aleman BMP, Raemaekers JMM, Tomsic R, et al.: Radiotherapy in advanced Hodgkin lymphoma (HL) patients in partial remission (PR) after chemotherapy: detailed results from the EORTC lymphoma group trial no.20884. [Abstract] Eur J Haematol 73 (Suppl 65): A-A01, 42, 2004.
- [Result] Aleman BM, Raemaekers JM, Henry-Amar M, et al.: Involved-field radiotherapy in patients with stage III/IV Hodgkin's lymphoma: first results of the randomised EORTC trial # 20884. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-3, 2, 2001.
- [Result] Raemaekers J, Burgers M, Henry-Amar M, Pinna A, Mandard A, Monfardini S, Hagenbeek A, Breed W, Carde P, Vovk M, van Hoof A, Thomas J, Noordijk E. Patients with stage III/IV Hodgkin's disease in partial remission after MOPP/ABV chemotherapy have excellent prognosis after additional involved-field radiotherapy: interim results from the ongoing EORTC-LCG and GPMC phase III trial. The EORTC Lymphoma Cooperative Group and Groupe Pierre-et-Marie-Curie. Ann Oncol. 1997;8 Suppl 1:111-4. PMID 9187443